CLINICAL TRIAL: NCT06648148
Title: Molecular Biomarkers of Response to Radiation Therapy in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other); University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: DCIS-2019
Record Dates: First submitted 2023-01-30; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify potential genetic and other molecular biomarkers of response to radiation therapy in breast cancer that may help to personalize breast cancer radiation treatment in the future.

DETAILED DESCRIPTION:
Monocentric prospective clinical study including DCIS patients treated at the Institute of Oncology Ljubljana. Patients treated with adjuvant radiotherapy and without systemic therapy are eligible for the study.

Adverse events of radiation treatment will be assessed after radiotherapy and during 5-year follow up and classified according to Common Terminology Criteria for Adverse Events v5.0.

Molecular biomarkers will be assessed before radiotherapy, after radiotherapy and during follow up. DNA will be isolated from whole blood samples obtained before radiation treatment. Circulating biomarkers will be isolated from plasma samples before treatment, after treatment and during follow-up. Written informed consent will be obtained from all included patients and the study design was approved by the National Medical Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with DCIS with an indication for adjuvant radiation therapy

Exclusion Criteria:

* Any specific systemic oncological therapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with non invasive ductal carcinoma in situ (DCIS) with an indication for postoperative radiation treatment.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events of radiation therapy | Within 1 month after completion of radiotherapy
  We will assess the proportion of patients exhibiting skin and cardiac adverse events after radiotherapy using Common Terminology Criteria for Adverse Events, NYHA class, measurement of cardiac biomarkers and cardiac imaging
Adverse events of radiation therapy | 6 months after radiotherapy
  We will assess the proportion of patients exhibiting skin and cardiac adverse events after radiotherapy using Common Terminology Criteria for Adverse Events, NYHA class, measurement of cardiac biomarkers and cardiac imaging
Adverse events of radiation therapy | 2 years after radiotherapy
  We will assess the proportion of patients exhibiting skin and cardiac adverse events after radiotherapy using Common Terminology Criteria for Adverse Events, NYHA class, measurement of cardiac biomarkers and cardiac imaging
Adverse events of radiation therapy | 5 years after radiotherapy
  We will assess the proportion of patients exhibiting skin and cardiac adverse events after radiotherapy using Common Terminology Criteria for Adverse Events, NYHA class, measurement of cardiac biomarkers and cardiac imaging

SECONDARY OUTCOMES:
Disease recurrence | 5 years after radiotherapy
  We will assess the proportion of patients with disease recurrence.
Disease recurrence | 10 years after radiotherapy
  We will assess the proportion of patients with disease recurrence.
Changes of circulating biomarkers | Within 1 month after completion of radiotherapy
  We will assess the changes of circulating biomarkers (miRNA, extracellular vesicles, proteins) after radiotherapy compared to values before radiotherapy.
Changes of circulating biomarkers | 6 months after radiotherapy,
  We will assess the changes of circulating biomarkers (miRNA, extracellular vesicles, proteins) after radiotherapy compared to values before radiotherapy.
Changes of circulating biomarkers | 2 years after radiotherapy
  We will assess the changes of circulating biomarkers (miRNA, extracellular vesicles, proteins) after radiotherapy compared to values before radiotherapy.
Changes of circulating biomarkers | 5 years after radiotherapy
  We will assess the changes of circulating biomarkers (miRNA, extracellular vesicles, proteins) after radiotherapy compared to values before radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Marinko, MD, PhD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No